CLINICAL TRIAL: NCT04715802
Title: Options of Breast Reconstruction Timing and Method After Removing of Polyacrylamide Hydrogel: a Propensity Score-matched Study
Brief Title: Options on the Breast Reconstruction Timing and Method After Removal of Polyacrylamide Hydrogel
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT20200748A
Record Dates: First submitted 2021-01-10; First posted 2021-01-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast; Mammaplasty; Breast Reconstruction
Keywords: polyacrylamide hydrogel (PAAG)
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- PAAG removal + Immediate implant reconstruction: Patients who had a one-stage operation comprising gel removal and immediate breast reconstruction.
  Interventions: Procedure: Immediate breast reconstruction with implant
- PAAG removal + Delayed implant reconstruction: Patients who had a two-stage operation comprising gel removal and delayed breast reconstruction at least 3 months later. The first included maximal gel removal and purulent tissue debridement, if necessary. Thereafter, patients were invited for a clinical follow-up and discussion about DBR 3 months later. The latter was offered as a second stage in those opting for it.
  Interventions: Procedure: delayed breast reconstruction with implant
- PAAG removal + No breast reconstruction: Patients who only underwent surgical PAAG removal without breast reconstruction.
- PAAG removal + Delayed autologous fat grafting reconstruction: Patients who underwent a two-stage operation comprising surgical PAAG removal and autologous fat injection at least 3months later. Usually, the amount of transplanted fat was 150-200mL/side. A multilayer and multi-tunnel injection method was commonly used.
  Interventions: Procedure: delayed breast reconstruction with autologous fat transplantation
- PAAG removal + breast reconstruction with implants: Patients who underwent surgical PAAG removal with immediate or delayed implant breast reconstruction.
- Primary breast augmentation with implants: Patients who had undergone conventional breast augmentation(BA) with implants during the study period who matched the study cohort by age(±5 years).

INTERVENTIONS:
Procedure: Immediate breast reconstruction with implant — Because most fillers are under the mammary gland, it is better to place the prosthesis into the opening under the pectoralis major muscle, which avoids contact between the prosthesis and the residual hydrogel to reduce the chance of infection. If postoperative complications disappear and imaging shows no filler remnants after more than 3-month follow-up, secondary breast augmentation can be planned. For placement of the prosthesis, the plane under the pectoralis major is preferred, which avoids prosthesis contact with the residual hydrogel to thus reduce the chance of infection.
  Other Names: Breast-Q questionnaire
  Groups: PAAG removal + Immediate implant reconstruction
Procedure: delayed breast reconstruction with implant — The first stage included maximal gel removal and purulent tissue debridement, if necessary. Thereafter, patients were invited for a clinical follow-up and discussion about DBR 3 months later. The latter was offered as a second stage in those opting for it.
  Other Names: Breast-Q questionnaire
  Groups: PAAG removal + Delayed implant reconstruction
Procedure: delayed breast reconstruction with autologous fat transplantation — Because fat injection after PAAG removal has a high infection risk, it is recommended to be conducted after 3-6 months of follow-up. The advantage of autologous fat transplantation is its ability to repair a variety of breast shape deformities caused by PAAG removal. Fat injections may need to be repeated several times. The interval between injections should be at least 3 months. Usually, the amount of transplanted fat is 150-200 mL/side. A multilayer and multi-tunnel injection method is commonly used.
  Other Names: Breast-Q questionnaireBreast-Q questionnaire
  Groups: PAAG removal + Delayed autologous fat grafting reconstruction

SUMMARY:
Since polyacrylamide hydrogel (PAAG) was used in cosmetic surgery in 1997, about 30 million women have received PAAG injection for breast augmentation. Although the use of PAAG has been prohibited in most countries due to its myriad complications, a large number of symptomatic patients and asymptomatic patients have continued to seek medical advice. The strategy of repairing secondary breast deformities after PAAG removal has increasingly become a concern for both doctors and patients, but there is no standardized algorithm yet. The purpose of the present study was to perform a retrospective study to compare the safety and effectiveness of different reconstruction timing and method after removing the gel.

DETAILED DESCRIPTION:
The primary purposes of this study are to:

1. Compare the safety and effectiveness of IBR vs DBR after PAAG removal;
2. Compare the safety and effectiveness of breast implants with silicone gel prosthesis vs autologous fat transplantation after PAAG removal;
3. Evaluate the clinical characteristics associated with and rates of complications based on reconstruction timing and type.

The secondary purposes of this study are to：

1. Explore and summarize the characteristics of long-term complications of PAAG injection for breast augmentation;
2. Compare the rate of postoperative complications and reoperations between the patients who had breast reconstruction with implants and patients who had primary breast augmentation with implants.
3. Further refine the algorithm for breast reconstruction in patients with PAAG injections.

ELIGIBILITY:
Inclusion Criteria:

1. history of PAAG breast injection;
2. appeal to remove the gel;
3. availability of complete medical records;
4. accepting the potential complications of the operation and breast deformity after gel removal.
5. agreeing with medical history data collection, clinical follow-up investigation, and independent Complete the questionnaire.

Exclusion Criteria:

1. Patients who had other breast diseases;
2. Patients who failed to follow the standard diagnosis, treatment and follow-up;
3. Lost to follow-up due to various reasons or incomplete medical records;
4. Patients with cognitive disorders such as mental illness, understanding, memory, or orientation, and other serious diseases.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who were admitted to the Plastic Surgery Department of the First Affiliated Hospital of Zhejiang University School of Medicine with complications after receiving PAAG injection for breast augmentation.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2006-10-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the occurrence of a postoperative complication | until 10 years post operation
  Complications are defined as any adverse postoperative events directly related to gel removal or breast reconstruction surgery that require further treatment. According to the patient's main complaint, physical examination, chest radiography, breast ultrasound, breast mammography or MRI, pathological biopsy and other methods to evaluate the complications. According to the degree of complications, they were further divided into: (1) Mild complications: conservative treatment without surgical treatment. (2) Severe complications: the incidence of complications requiring reoperations or implant removal/replacement operations.
The probability of reoperations | until 10 years post operation
  Reoperation was defined as a surgical event performed after PAAG removal alone or stage I and II reconstruction. An anticipated operation of delayed breast implantation in patients with two-stage surgery was not classified as reoperation.

SECONDARY OUTCOMES:
Patient-reported quality of life, QOL | until 1 year post operation
  Patient-reported quality of life using Breast-Q score to evaluate changes in breast appearance, mental health, physical health and sexual health satisfaction before and after surgery.
Aesthetic evaluation | until 1 year post operation
  It was evaluated by the Aesthetic Items Scale, which was a standardized tool for evaluating the aesthetic effect of breast reconstruction surgery, which was first proposed by Visser and Brinkman. The specific method was as follows: 3 experienced plastic surgeons evaluate 5 standardized photos (front, oblique, and side) of the patient before and after surgery. All photos were organized into slides and displayed randomly, with other information hidden (Such as preoperative or postoperative state, reconstruction method used, complications or whether to perform a second operation, etc.). In order to minimize the deviation, blank slides were displayed between the photos, and the random order of the photos of each observer was different. Each doctor used a five-point Likert scale to score breast volume, shape, symmetry, scars, and nipple areola. In addition, each doctor gave an overall satisfaction score between 0-10 points based on pre- and post-operative photos.
change in patient satisfaction | until 1 year post operation
  Patient satisfaction consisted of four structured questions that assessed satisfaction with the size, shape, symmetry, and sensitivity of the breast. Patients were asked to rate their final result as "good", "satisfactory", "poor" or "bad".

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Plastic and Reconstructive Surgery, The First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China